CLINICAL TRIAL: NCT01195987
Title: Immune Dysregulation in Hepatitis C Patients With or Without Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Center for Rheumatic Disease, Allergy, & Immunology (Other)
Collaborators: St. Luke's Hospital (Unknown)
Responsible Party: Dr. Nabih I Abdou, PhD, Center for Rheumatic Disease, Allergy, & Immunology
Other Study IDs: 09-290
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Hepatitis C Patients
Keywords: Hepatitis C; Arthritis
MeSH Terms: conditions — Hepatitis C; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hepatitis C with Arthritis
- Hepatitis C without Arthritis

SUMMARY:
The purpose of this study is to study the role of the Immune System in causing arthritis in patients with Hepatitis C.

DETAILED DESCRIPTION:
Patients will provide one blood sample after qualifying for the study, and signing consent. The patients will have a skin test TB, Candida, and Trichophyton placed and will read the results themselves and mail back the card with the measurements to be recorded. Labs will test for ESR, CBC, CRP, antiCCP, Cryoglobulins, RF, CH50, C3, C4, Flow cytometry, and would have already been tested for HIV and Hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* All adults 18 or older, 20 will have hep C positive with a viral load withen 6 mo. of enrollment.
* Either interferon or antiviral naive or those who failed interferon or antiviral therapy more than 6 mo. prior to enrollment.
* 10 normal healthy controls- Hep C neg and without osteoarthritis (OA).

Exclusion Criteria:

* HIV patients
* Those with concomitant alcoholic liver disease
* Patients with Rheumatoid Arthritis (RA) or other autoimmune disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hepatitis positive patients with and without osteoarthritis, with a group of Hepatitis C negative and no osteoarthritis to serve as controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nabih I Abdou, MD, PhD, Principal Investigator — Center for Rheumatic Disease, Allergy & Immunology
Locations (1):
- Center for Rheumatic Disease, Allergy & Immunology, Kansas City, Missouri, United States